CLINICAL TRIAL: NCT00529113
Title: A Randomized Phase I/II Study With Gemcitabine and RTA 402 or Gemcitabine and Placebo for Patients With Unresectable Pancreatic Cancer
Brief Title: Study With Gemcitabine and RTA 402 for Patients With Unresectable Pancreatic Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: To pursue other indications
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 402-C-0702
Record Dates: First submitted 2007-09-12; First posted 2007-09-14 (Estimated); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Pancreatic Neoplasms; Pancreatic Cancer
Keywords: pancreatic cancer; gemcitabine
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — bardoxolone methyl; Gemcitabine

ARMS (9):
- Phase 1 Cohort 1 (Experimental): Bardoxolone methyl 150 mg/day x 21 days and gemcitabine (1000 mg/m2 by intravenous infusion on Days 1, 9, and 15)
  Interventions: Drug: Bardoxolone methyl; Drug: Gemcitabine
- Phase 1 Cohort 2 (Experimental): Bardoxolone methyl 300 mg /day for 21 days and gemcitabine (1000 mg/m2 by intravenous infusion on Days 1, 9, and 15)
  Interventions: Drug: Bardoxolone methyl; Drug: Gemcitabine
- Phase 1 Cohort 3 (Experimental): Bardoxolone methyl 150 mg/day for 28 days and gemcitabine (1000 mg/m2 by intravenous infusion on Days 1, 9, and 15)
  Interventions: Drug: Bardoxolone methyl; Drug: Gemcitabine
- Phase 1 Cohort 4 (Experimental): Bardoxolone methyl 200 mg/day for 28 days and gemcitabine (1000 mg/m2 by intravenous infusion on Days 1, 9, and 15)
  Interventions: Drug: Bardoxolone methyl; Drug: Gemcitabine
- Phase 1 Cohort 5 (Experimental): Bardoxolone methyl 250 mg/day for 28 days and gemcitabine (1000 mg/m2 by intravenous infusion on Days 1, 9, and 15)
  Interventions: Drug: Bardoxolone methyl; Drug: Gemcitabine
- Phase 1 Cohort 6 (Experimental): Bardoxolone methyl 300 mg/day x 28 days and gemcitabine (1000 mg/m2 by intravenous infusion on Days 1, 9, and 15)
  Interventions: Drug: Bardoxolone methyl; Drug: Gemcitabine
- Phase 1 Cohort 7 (Experimental): Bardoxolone methyl 350 mg/day x 28 days and gemcitabine (1000 mg/m2 by intravenous infusion on Days 1, 9, and 15)
  Interventions: Drug: Bardoxolone methyl; Drug: Gemcitabine
- Phase 2 Cohort 1 (Experimental): Bardoxolone methyl maximum tolerated dose(as determined in the Phase 1 portion of the study)/day x 28 days and gemcitabine (1000 mg/m2 by intravenous infusion on Days 1, 9, and 15)
  Interventions: Drug: Gemcitabine; Drug: Bardoxolone methyl
- Phase 2 Cohort 2 (Placebo Comparator): Placebo capsules/day x 28 days and gemcitabine (1000 mg/m2 by intravenous infusion on Days 1, 9, and 15)
  Interventions: Drug: Gemcitabine; Drug: Placebo

INTERVENTIONS:
Drug: Bardoxolone methyl — Bardoxolone methyl capsules (150 mg/day) for 21 days
  Other Names: RTA 402
  Arms: Phase 1 Cohort 1
Drug: Bardoxolone methyl — Bardoxolone methyl capsules (300 mg/day) for 21 days
  Other Names: RTA 402
  Arms: Phase 1 Cohort 2
Drug: Bardoxolone methyl — Bardoxolone methyl capsules (150 mg/day) for 28 days
  Other Names: RTA 402
  Arms: Phase 1 Cohort 3
Drug: Bardoxolone methyl — Bardoxolone methyl capsules (200 mg/day) for 28 days
  Other Names: RTA 402
  Arms: Phase 1 Cohort 4
Drug: Bardoxolone methyl — Bardoxolone methyl capsules (250 mg/day) for 28 days
  Other Names: RTA 402
  Arms: Phase 1 Cohort 5
Drug: Bardoxolone methyl — Bardoxlone methyl capsules (300 mg/day) x 28 days
  Other Names: RTA 402
  Arms: Phase 1 Cohort 6
Drug: Bardoxolone methyl — Bardoxolone methyl capsules (350 mg/day) x 28 days
  Other Names: RTA 402
  Arms: Phase 1 Cohort 7
Drug: Gemcitabine — 1,000 mg/m2 administered as an intravenous infusion on days 1, 8, and 15
  Other Names: Gemzar
Drug: Placebo — Placebo capsules x 28 days
  Arms: Phase 2 Cohort 2
Drug: Bardoxolone methyl — Bardoxolone methyl maximum tolerated dose (as determined in the Phase 1 portion of the study)/day x 28 days
  Other Names: RTA 402
  Arms: Phase 2 Cohort 1

SUMMARY:
This study assesses the safety and efficacy of RTA 402 in combination with gemcitabine in patients with unresectable pancreatic cancer.

DETAILED DESCRIPTION:
Phase I will be conducted to determine the MTD of RTA 402 (administered orally Days 1-21 or Days 1-28 of a 28-day cycle) in combination with gemcitabine (1000 m/m2). Gemcitabine will be administered as an intravenous infusion on Days 1, 8, and 15 of each 28-day cycle.

The phase II portion of the study will be randomized, and double-blinded. Phase II will utilize the RTA 402 MTD determined in Phase I; Arm 1 will consist of gemcitabine + RTA 402. RTA 402 capsules will administered orally Days 1-21 of each 28-day cycle (or Days 1-28 if appropriate, based on phase I results); gemcitabine (1000 mg/m2) will be administered as an intravenous infusion on Days 1, 8, and 15 of each 28-day cycle in each Arm. Arm 2 will consist of gemcitabine + placebo, placebo capsules will be taken orally Days 1-21 of each 28-day cycle (or Days 1-28 if appropriate, based on phase I results). Both treatment arms are 4-weeks in length.

The study was conceived with both a Phase I and Phase II portion as described above; however, only the Phase I portion was completed. The trial was terminated in 2009 before the Phase II portion could begin.

ELIGIBILITY:
Inclusion Criteria:

* Phase I patients should have treatment naïve pancreatic cancer; however , Phase I patients who have had 1 prior regimen consisting of adjuvant chemo-radiation or adjuvant gemcitabine - as defined within the NCCN guidelines may be enrolled. Phase II patients must have metastatic disease (Stage IV only).
* Karnofsky performance status of >70%
* Adequate liver function. (total bilirubin ≤ 1.5 mg/dL and AST(SGOT) and ALT(SGPT) of < 2.5 ULN ( ≤ 5 ULN for Phase II patients with liver metastases), Serum Creatinine < 1.5 ULN
* Adequate bone marrow function as documented by the following laboratory test results within 14 days of starting therapy. platelets ≥100,000/mm3, absolute neutrophil count (ANC) ≥1500/mm3, hemoglobin ≥9.0 g/dL, white blood cell (WBC) count ≥3000 /mm3
* Practice effective contraception during the entire study period.
* Life expectancy of more than 3 months.
* Able and willing to sign the informed consent form.
* Willing and able to self-administer orally and document all doses of RTA 402 ingested.

Exclusion Criteria:

* Prior treatment for current malignancy outside of the adjuvant setting for Phase I
* Inability to swallow tablets or capsules
* Active brain metastases or primary central nervous system (CNS) malignancies. (Patients with a previously treated brain metastasis may be included.)
* Active second malignancy
* Ten percent or greater weight loss over the 6 weeks before study entry.
* Pregnant or breast feeding
* Clinically significant illnesses which could compromise participation in the study, including, but not limited to: Uncontrolled diabetes; Active or uncontrolled infection; Acute or chronic liver disease; Confirmed diagnosis of Human immunodeficiency virus (HIV) infection; Uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction within the past 6 months, or uncontrolled cardiac arrhythmia.
* Psychiatric illness that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2007-09-30 (Actual); Primary Completion 2009-11-01 (Actual); Study Completion 2009-11-01 (Actual)

PRIMARY OUTCOMES:
Phase I - To determine the maximum tolerated dose (MTD) of RTA 402 in combination with gemcitabine in patients with locally advanced or metastatic pancreatic cancer. | End of trial
Phase II - To determine if treatment with RTA 402 in combination with gemcitabine can increase the progression-free survival versus gemcitabine plus placebo in patients with unresectable metastatic pancreatic cancer. | End of Trial

SECONDARY OUTCOMES:
Phase I - To document any preliminary antitumor activity of RTA 402 in this patient population. | End ofTrial
Phase I - To characterize the pharmacokinetics (PK) of RTA 402 in this population. | End of Trial
Phase II - To determine the overall response rate in patients treated with RTA 402 + gemcitabine and in patients treated with gemcitabine + placebo. | End of Trial
Phase II - To determine the 1-year survival in this patient population. | End of Trial
Phase II - To determine the toxicities of these regimens. | End of Trial
Phase II - To determine the changes in quality of life (Functional Assessment of Chronic Illness Therapy (Fatigue), [FACIT-F]). | End of Trial

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Rocky Mountain Cancer Center (US Oncology), Denver, Colorado
  - Cancer Centers of Florida (US Oncology), Ocoee, Florida
  - Central Indiana Cancer Centers (US Oncology), Indianapolis, Indiana
  - Sammons Cancer Center (US Oncology), Dallas, Texas
  - Northwest Cancer Specialist- Vancouver Cancer Specialist (US Oncology), Vancouver, Washington

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/